CLINICAL TRIAL: NCT05303558
Title: Real World Outcome Analysis for APAC High Risk Localized Prostate Cancer Patients Treated With Radical Prostatectomy and Perioperative Hormonal Therapy
Brief Title: A Study of High Risk Localized Prostate Cancer Participants Treated With Radical Prostatectomy and Perioperative Hormonal Therapy
Acronym: ACE
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson International (Singapore) Pte. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109188; NOPRODPCR4002 (Other: Johnson & Johnson International (Singapore) Pte Ltd)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: High Risk Localized Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With High-risk Localized Prostate Cancer: Adult participants from Japan, South Korea, and Taiwan with high-risk localized prostate cancer (HR LPC) who received radical prostatectomy (RP) and perioperative (neoadjuvant and/ or adjuvant) hormonal therapy will be observed from the date of confirmed HR LPC diagnosis until death, lost to follow-up (last known visit), or end of study period, whichever comes first. This study will utilize data from electronic medical records (EMR) in South Korea and Taiwan, and data from chart reviews in Japan. Data will be analyzed retrospectively from 1 January 2015 to 30 June 2017, with a follow-up till 30 June 2022.

SUMMARY:
The purpose of this study is to evaluate the yearly conditional prostate-specific antigen (PSA) progression-free survival (PFS) probabilities in high-risk localized prostate cancer (HR LPC) participants following radical prostatectomy (RP) and perioperative hormonal therapies (that is, hormonal treatment before RP and / or after RP) over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have histologically confirmed adenocarcinoma of the prostate
* Participants newly diagnosed between 1 January 2015 to 30 June 2017 (both dates inclusive)
* Participants fulfil high-risk localized prostate cancer defined by national comprehensive cancer network (NCCN) prostate cancer guideline (2020 version 1) a. T3a or; b. Grade group 4 or Grade group 5 or; c. Prostate specific antigen (PSA) greater than (>) 20 nanograms per milliliter (ng/mL)
* Participants must have received radical prostatectomy (RP) between 1 January 2015 and 30 June 2017
* Participants must have received at least one perioperative hormonal therapy pattern as listed below:

  1. greater than or equal to (>=) 3 months neoadjuvant hormonal therapy, duration between date of last dose and date of RP should be less than or equal to (<=) 2 months; and/or
  2. >= 6 months adjuvant hormonal therapy, first dose started within 6 months of RP surgery

     Exclusion Criteria:
* Distant metastasis based on conventional imaging (clinical stage M1) at time of prostate cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes newly diagnosed adult high-risk localized prostate cancer (HR LPC) participants who received radical prostatectomy (RP) and perioperative hormonal therapy.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Yearly Conditional Prostate-specific Antigen (PSA) Progression-free Survival (PFS) Probability | Up to 5 years
  PSA PFS probability is defined as probability of being PSA progression free given that participant has yet to experience PSA progression or death from any cause. PSA progression is defined as per the prostate cancer working group 2 (PCWG2) consensus.

SECONDARY OUTCOMES:
Localized Prostate Cancer (LPC) Stage at Diagnosis | Up to 2.5 years
  LPC stage at diagnosis will be based on the latest tumor nodes and metastases (TNM) staging system approved by the American Joint Committee on Cancer (AJCC).
Time from Diagnosis of LPC to Radical Prostatectomy (RP) | Up to 2.5 years
  Time from diagnosis of LPC to RP will be reported.
Number of Participants who Received Treatments Provided with RP and Following RP | Up to 7.5 years
  Number of participants who received treatments provided with RP and following RP (including RP and neo-adjuvant hormonal therapy only, RP and adjuvant hormonal therapy only, or RP and both neoadjuvant and adjuvant hormonal therapies) will be reported.
Hormonal Therapy Duration | Up to 7.5 years
  Hormonal therapy duration is defined as the length of time between the start date of receiving hormonal therapy treatment and the date of receiving last dose.
Yearly Conditional Local or Distant Radiographic PFS Probability | Up to 5 years
  Conditional radiographic PFS probability is defined as the probability of being radiographic progression-free given that participant has yet to experience local or distant radiographic progression.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson International (Singapore) Pte Ltd Clinical Trial, Study Director — Johnson & Johnson International (Singapore) Pte. Ltd.
Locations (9):
- Japan (5):
  - Akita University Hospital, Akita
  - Hirosaki University Hospital, Hirosaki
  - Nagoya City University Hospital, Nagoya
  - Yokohama City University Hospital, Yokohama
  - Yokosuka Kyosai Hospital, Yokosuka
- South Korea (3):
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Catholic Medical Center, Seoul
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No